CLINICAL TRIAL: NCT05722444
Title: Investigation of Sleep and Health Outcomes in Women Reporting Heavy Menses Flow
Brief Title: Sleep and Health Outcomes in Women With Heavy Menses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jessica Walter, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00215465
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Menstruation; Heavy
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with reported heavy menses (Experimental)
  Interventions: Other: Nighttime Feminine Product

INTERVENTIONS:
Other: Nighttime Feminine Product — During nights while menstruating:
  * Standardized nighttime feminine product + typical nighttime behaviors to prevent leak
  * Standardized nighttime feminine product + refraining from nighttime behaviors to prevent leak

SUMMARY:
This study will evaluate subjective sleep over three consecutive menstrual cycles (menses and non-menses) in females reporting heavy menstrual bleeding. Following a baseline phase of one menstrual cycle, study subjects will use a standardized nighttime feminine product during menstruation for their second cycle. For the third cycle, subjects will continue to use the standardized menstrual product with behavioral modification that includes refraining from those sleep behaviors used to avoid nighttime menstrual leakage.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50 years old
* Generally healthy (self-assessed; no significant underlying disease)
* Premenopausal patients with regular menstrual cycles every 21 to 35 days
* Patients with at least 3 days and no more than 7 days of bleeding during menstruation
* An intact uterus and at least one ovary
* Ability and willingness to provide written informed consent
* Willingness to adhere to study procedures
* Menstrual pads are the primary form for nighttime menstrual protection needs
* Will maintain a daily schedule that allows normal or typical sleep habits (ie, not a night-shift worker; >5 hours of sleep).
* Women will self-report that they have heavy flow and perform at least one of the following compensatory behaviors:

  * Set an alarm or plan to get up in the middle of the night to check or change the pad
  * Add additional disposable absorbent products for extra leak protection of coverage (e.g. extra pads or liners)
  * Use pillows or other means to limit sleep positions (to prevent moving at night)
  * Use something extra on top of my bedding (such as a towel) to sleep on
  * Wear an extra pair of pants/shorts
  * Wear tighter clothing than they typically would, like yoga pants

Exclusion Criteria:

* Currently pregnant or intending to imminently attempt pregnancy
* Any condition (social or medical) that, in the opinion of the primary care giver or study staff, would make trial participation unsafe or complicate data interpretation
* Difficult sleeping environment due to:

  * Frequently involved in activities requiring nighttime awakenings (eg, taking care of an infant or loved one).
  * Disruptive bed partners (i.e., snoring, children, pets, etc)
  * Diagnosed sleep disorders (i.e. insomnia, sleep apnea, restless leg disorder, breathing disorder, etc)
* Use of an Intrauterine Device (IUDs) unless copper IUD.
* Regular use (>1 day per week) of sleep aids and/or sedating medications, including over the counter products like melatonin.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants who are born female/undergoing menstruation.
Enrollment: 25 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | 3 months
  Determine the change in PSQI over the 3 months of study participation. Maximum score is 21 (worse sleep outcomes) and minimum score is 0 (better sleep outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States